CLINICAL TRIAL: NCT03735095
Title: Endobronchial Ultrasound Transbronchial Needle Guided Interstitial Photodynamic Therapy for Palliation of Locally Advanced Lung Cancer and Advanced Cancers Obstructing the Airway -Phase I/II
Brief Title: Endobronchial Ultrasound Guided Interstitial Photodynamic Therapy in Treating Patients With Locally Advanced Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: was paused by device company for a long period of time
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pinnacle Biologics Inc. (Industry); Simphotek Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 279415; NCI-2018-01969 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 279415 (Other: Roswell Park Cancer Institute); 1R44CA265656 (NIH)
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Lung Carcinoma; Non-Small Cell Lung Carcinoma; Small Cell Lung Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (porfimer sodium, EBUS, and photodynamic therapy) (Experimental): Treatment (porfimer sodium, EBUS, and photodynamic therapy) Patients receive 2 mg/kg porfimer sodium IV over 3-5 minutes 48 +/- 4 hours prior to the delivery of I-PDT. Patients then undergo EBUS-TBN guided I-PDT over few hours.
  Interventions: Drug: Porfimer Sodium; Procedure: Ultrasound-Guided Transbronchial Needle-Delivered Interstitial Photodynamic Therapy

INTERVENTIONS:
Drug: Porfimer Sodium — Given IV
  Other Names: Photofrin
Procedure: Ultrasound-Guided Transbronchial Needle-Delivered Interstitial Photodynamic Therapy — Undergo EBUS-TBN guided I-PDT
  Other Names: Endobronchial Ultrasound with Transbronchial Needle (EBUS-TBN) Guided Interstitial PDT (IPDT); Endobronchial Ultrasound Transbronchial Needle-Guided Interstitial Photodynamic Therapy; Ultrasound-Guided Transbronchial Needle-Guided Interstitial Photodynamic Therapy; EBUS-TBN Interstitial Photodynamic Therapy; EBUS-TBN IPDT

SUMMARY:
This Phase I/Il studies the side effects of endobronchial ultrasound guided interstitial photodynamic therapy work in treating patients with lung cancer that has spread to nearby tissues or lymph nodes. Photodynamic therapy consists of injecting a light sensitive drug called a photosensitizer, such as porfimer sodium, into the vein, waiting for it to accumulate in the tumor, and then activating it with a red laser light. Giving photodynamic therapy with Porfimer sodium may reduce the tumor size in patients with lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES PHASE 1:

I. To evaluate the safety and potential efficacy of endobronchial ultrasound with transbronchial needle (EBUS-TBN) guided interstitial photodynamic therapy (EBUS-TBN I-PDT) and/or I-PDT and/or photodynamic therapy (PDT) in patients with malignant airway obstructions using porfimer sodium as a photosensitizer.

PRIMARY OBJECTIVE Phase II

* I. To assess the tumor response to treatment.
* II To observe changes in well being

SECONDARY OBJECTIVES:

* I. To evaluate local progression-free survival (PFS).
* II.To compare the treatment planning in DOSIE™ with the plan generated in COMSOL™ - COHORT A ONLY
* III. To measure changes in tumor pO2, optical properties, and irradiance and fluence in relationship to response

EXPLORATORY OBJECTIVES:

I. Examine porfimer sodium retention in the target tumor tissue. II. Examine the relationship between immune biomarkers and response.

OUTLINE:

Patients receive Porfimer sodium intravenously (IV) over 20 minutes delivery of I-PDT. 20 minutes 48 hours +/- 4 hours before receiving I-PDT. I-PDT is then received over 1-2 hours.

After completion of study treatment, patients are followed up at 4, 8, 12, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* > 18 year olds
* Eligibility checklist before registration requires review of case by study surgeon or interventional pulmonologists to approve anatomic feasibility of an airway intervention
* For patients in Cohort B only. Patients are amenable to receive a palliative radiotherapy of 8 Gy x1 48±4 h prior to the I-PDT, as determined by the radiation oncologist
* Patients with an established pathologic diagnosis of small cell and/or non-small cell lung cancer or other malignancies causing airway obstruction > 25% requiring bronchoscopic intervention. Or inoperable malignancies not candidates for curative radiotherapy within the airway.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 3
* Platelets >= 100,000 cells/mm^3 (International System of Units [SI] units 100 x 10^9/L).
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Participants who have had radiotherapy to the target tumor within 4 weeks prior to the scheduled I-PDT and/or PDT.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing female participants.
* Co-existing ophthalmic disease likely to require slit-lamp examination within 14 days following I-PDT and/or PDT treatment.
* Known hypersensitivity/allergy to porphyrin.
* Patients who are not cleared by the anesthesiologist to undergo an advanced bronchoscopy procedure under general anesthesia.
* Patients with target tumor invading into the lumen of the esophagus, confirmed by esophago-gastro-duodenoscopy (EGD) with endoscopic ultrasound
* Patients diagnosed with porphyria.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive I-PDT or PDT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Ivanick, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Porfimer Sodium, EBUS, and Photodynamic Therapy): Patients received IV of 2 mg/kg porfimer sodium over 3-5 minutes and 48 hours +/- 4 prior the I-PDT. Patients then undergo EBUS-TBN guided I-PDT over a few hours.
  Porfimer Sodium: Given IV Ultrasound-Guided Transbronchial Needle-Delivered Interstitial Photodynamic Therapy: Undergo EBUS-TBN guided I-PDT Interstitial Photodynamic Therapy: Undergo EBUS-TBN guided I-PDT
Period: Overall Study
Arm/Group | Treatment (Porfimer Sodium, EBUS, and Photodynamic Therapy)
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Treatment (Porfimer Sodium, EBUS, and Photodynamic Therapy): Patients received IV of 2 mg/kg porfimer sodium over 3-5 minutes and 48 hours +/- 4 prior the I-PDT. Patients then undergo EBUS-TBN guided I-PDT over a few hours.
  Porfimer Sodium: Given IV Ultrasound-Guided Transbronchial Needle-Delivered Interstitial Photodynamic Therapy: Undergo EBUS-TBN guided I-PDT
Arm/Group | Treatment (Porfimer Sodium, EBUS, and Photodynamic Therapy)
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events That Are >= Grade 4 According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.0
Description: Number of Participants with Adverse Events That Are >= Grade 4 According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.0
Time Frame: Up to 4 weeks
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Porfimer Sodium, EBUS, and Photodynamic Therapy)
Number analyzed (Participants) | 19
Participants | 6

2. Primary Outcome: Number of Participants With Tumor Response
Description: Will be reported using frequencies
Time Frame: up to 24 weeks
Population: All treated and eligible patients
Measure: Number; unit: participants
Arm/Group | Treatment (Porfimer Sodium, EBUS, and Photodynamic Therapy)
Number analyzed (Participants) | 19
participants | 0

3. Secondary Outcome: Progression-free Survival (PFS) Assessed Using Modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Criteria
Description: Will be summarized using standard Kaplan-Meier methods, with median progression-free survival (PFS) estimated with 95% confidence intervals.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From initiation of treatment to time of first observed diseased progression or death assessed up to 24 weeks
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Porfimer Sodium, EBUS, and Photodynamic Therapy)
Number analyzed (Participants) | 19
months | 2.6 [0.9 to 5.9]

ADVERSE EVENTS:
Time Frame: Up to 4 months
Arm/Group | Treatment (Porfimer Sodium, EBUS, and Photodynamic Therapy)
All-Cause Mortality (participants affected / at risk) | 17/19
Serious Adverse Events (participants affected / at risk) | 12/19
Other Adverse Events (participants affected / at risk) | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Porfimer Sodium, EBUS, and Photodynamic Therapy) (N=19)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Esophageal fistula (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (3)
Platelet count decreased (Investigations) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Porfimer Sodium, EBUS, and Photodynamic Therapy) (N=19)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Esophageal fistula (Gastrointestinal disorders) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 4 (5)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (6)
Fever (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4)
Pain (General disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Cardiac troponin T increased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03735095/Prot_SAP_000.pdf